CLINICAL TRIAL: NCT05399433
Title: Rôle du métabolisme du Glucose Dans la Migration Des Cellules Dendritiques cutanées Dans le Psoriasis : étude Pilote Translationnelle
Brief Title: Role of Glucose Metabolism in Migration of Cutaneous Dendritic Cells in Psoriasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-PP-25
Record Dates: First submitted 2022-05-16; First posted 2022-06-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Production of IL-23 of blood and skin dendriti cells (CD) (Other): Simultaneously evaluate the migratory capacity and production of IL-23 of blood and skin cDC on peripheral venous blood and skin biopsies of psoriatic patients with and without type 2 diabetes and control patients (with or without type II diabetes) depending on their metabolic status.
  Interventions: Other: Biopsy and venous blood

INTERVENTIONS:
Other: Biopsy and venous blood — A skin biopsy will be performed under local anesthesia in diabetic and non-diabetic psoriatic patients (25 per group) in the injured area (joint extension) and in the non-injured area more than 2 cm from any lesion in the same area. In patients in the diabetic or non-diabetic control group (25 per group) only one biopsy will be performed.
  Peripheral venous blood will be collected in heparin tubes for metabolic parameter analysis and blood CD analysis

SUMMARY:
Dendritic cells (DC) paly a key role in the induction and chronicity of psoriasis by capturing the antigenes and activating the T cell repsonse. This activation requires their migration from the cutaneous sensitisation site to the lymph nodes. This migration requires an important intracellular metabolic activity, with a strong involvmenet of glucdic metabolism. This activity is linked with the systemic activity. This study aims to compare the migration and the phenotypic and metabolic caracteristics of blood and skin DCs in patients with or without psoriasis and with or without type 2 diabetes,

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* hospitalized in the Dermatology department of the CHU of Nice for moderate to severe psoriasis (defined by a PASI > or = 10)
* covered by a social security scheme after obtaining a free
* Clinical diagnosis of plaque psoriasis by a dermatologist with or without type 2 diabetes (defined by glycated hemoglobin >7%)
* For the control group: without psoriasis or other inflammatory dermatosis aged in the presence or not of type 2 diabetes (glycated hemoglobin >7%).
* free and informed consent

Exclusion Criteria:

* Minor or incapable or unwilling to consent freely or in an informed manner Pregnant or nursing woman.
* Patient in a period of exclusion from other biomedical research
* Patient with generalized chronic inflammatory disease or other inflammatory dermatosis
* Patients on general corticosteroid, immunomodulator or immunosuppressant therapy in the month prior to local inclusion or treatment with corticosteroid therapy in the 15 days prior to inclusion, on anti- treatmentIL-23 or anti IL12/23 for less than 3 months or under anti-IL-17 or anti-TNF treatment for less than 1 month.
* Contraindication to cutaneous biospsis (known hemostasis disorder, taking anticoagulants, allergy to xylocaine, history of cheloid scars, congenital immune deficiency)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of dentridic cells producers of IL-23 | at baseline
  Alterations in the percentage of dentridic cells that have migrated with the metabolic status of patients

SECONDARY OUTCOMES:
Percentage of subpopulations dentridic cells producers | At baseline
  Study of the percentage of the various cDC subpopulations according to the metabolic status of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: passeron thierry, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France